# INVITATION TO PARTICIPATE IN THE RESEARCH PROJECT

# EMOTION REGULATION SKILLS TRAINING AND TRAUMA-FOCUSED THERAPY IN TREATMENT FOR SUBSTANCE USE DISORDER

### Molde Treatment Center 2021-2026

Many individuals with severe substance abuse struggle to cope with difficult emotions and have experienced serious traumas. Both factors have been shown to correlate with a higher likelihood of treatment disruption and relapse to substance use following treatment. In this study, we aim to investigate these relationships more closely, with a particular focus on feelings of shame, guilt, and emotional avoidance. In the study, we will address difficulties in managing emotions using a method called Dialectical Behavior Therapy (DBT). Patients with post-traumatic symptoms will also be offered the effective trauma therapy called Narrative Exposure Therapy (NET). We believe that this approach will result in fewer patients relapsing into substance use after completing treatment. You are being asked to participate in the study because you are admitted to treatment at Molde Treatment Center.

### WHAT DOES THE PROJECT ENTAIL?

In addition to regular psychological assessment, you will be specifically assessed for difficulties in managing difficult emotions and post-traumatic symptoms. This assessment will take place approximately 5 weeks after admission. Following this, you will be offered to participate in Dialectical Behavior Therapy (DBT) -skill training focusing on managing difficult emotions without the use of substances using. The start date will vary slightly in relation to other aspects of your treatment plan. This skill training will take place in groups of 6-8 patients over a period of 10 weeks. We will conduct two sessions per week, each lasting two hours. Here, you will learn practical skills to help you manage difficult emotions, increase here and now presence, crisis management, and maintain relationships with others. Those with post-traumatic symptoms will also be offered Narrative Exposure Therapy (NET). This will begin 1-2 weeks after you start the skill training. At the beginning of therapy, you will receive information and training on post-traumatic symptoms. Then, together with your therapist, you will create a lifeline where you briefly mention your traumatic experiences in addition to positive events and any instances where you have caused harm to others. Sessions will last for 90 minutes, and you will have 1-2 sessions per week for the same 10 weeks as the DBT treatment. During these sessions, you will go through the traumatic events in more detail with your therapist, with the aim of reducing the post-traumatic discomfort over time. Both of these treatment interventions will be in addition to the regular treatment provided at MBS. Four weeks after you have completed the treatment described above, we will assess the benefits of the treatment. Three and twelve months after discharge, we will contact you to conduct follow-up assessments to see how you are doing.

In the project, we will collect and record information about you. We will register slightly more information than usual in relation to psychological assessment, and we will also record information about the benefits of the treatment afterwards. We use interviews and questionnaires in addition to information from medical records.

### REASONABLE, EXPECTED RISKS AND BENEFITS

Participants in the project are likely to develop better skills in managing difficult emotions without using substances, and any potential post-traumatic symptoms are likely to improve. This will probably better equip you to remain abstinent from substances following treatment. Trauma therapy may initially cause some increased discomfort, such as increased anxiety. However, there is good evidence that symptoms improve throughout the course of treatment, and with good long-term effects. Research has shown that some individuals discontinue this type of trauma treatment when it is conducted outside the facility (outpatient). This may be due to the short-term increase in symptoms that some experience. Since we are addressing trauma concurrently with training on managing difficult emotions, we believe more patients will be able to complete treatment than is usual in substance abuse treatment.

### VOLUNTARY PARTICIPATION AND POSSIBILITY TO WITHDRAW CONSENT

Participation in the project is voluntary. If you wish to participate, you will sign the consent form on the last page. You may withdraw your consent at any time and without stating any reason. If you withdraw from the project, you may request that collected samples and information be deleted, unless the information has already been included in analyses or used in scientific publications. If you later wish to withdraw or have questions about the project, you can contact:

Medical Doctor Edvard Breivik. Email: edvard\_breivik@hotmail.com Phone: 93032613

Psychologist Johanna Vigfusdottir. Email: johannavigfusd@gmail.com Phone: 46746154

### WHAT HAPPENS TO THE INFORMATION ABOUT YOU?

The information recorded about you will only be used as described in the purpose of the project. You have the right to access the information recorded about you and the right to have any errors in the recorded information corrected. You also have the right to access the security measures regarding the processing of the information.

All information will be processed without names and national identification numbers or other directly identifiable information. A list with names and participant numbers is the only link between your information and your name. Only Edvard Breivik and Johanna Vigfusdottir have access to this list.

Information about you will be anonymized or deleted five years after the end of the project.

### **INSURANCE**

The Patient Injury Act will apply as usual.

# APPROVAL

The Regional Committee for Medical and Health Research Ethics has reviewed the project and has given preapproval (203 428/2020).

Under the new Personal Data Act, the data controller at the Molde Treatment Center and the project leader, Chief Physician Egil Jonsbu, have independent responsibility for ensuring that the processing of your information has a legal basis. This project has legal basis under the EU General Data Protection Regulation Article 6 no. 1a and Article 9 no. 2a and your consent.

You have the right to complain about the processing of your information to the Data Inspectorate.

# **CONTACT INFORMATION**

If you have any questions about the project, you can contact:

Medical Doctor Edvard Breivik. Email: <a href="mailto:edvard-breivik@hotmail.com">edvard-breivik@hotmail.com</a> Phone: 93032613

Psychologist Johanna Vigfusdottir. Email: <u>johannavigfusd@gmail.com</u> Phone: 46746154

The institution's data protection officer is <a href="mailto:personvernombud@helse-nordtrondelag.no">personvernombud@helse-nordtrondelag.no</a>

# I CONSENT TO PARTICIPATE IN THE PROJECT AND TO MY PERSONAL INFORMATION BEING USED AS DESCRIBED

| Date and place | Participant signature |
|----------------|---------------------------------------|
| | Participant name with capital letters |